CLINICAL TRIAL: NCT07328204
Title: Comprehensive Efficacy Study of Kasai Portoenterostomy for Biliary Atresia Stratified by Refined Surgical Timing: A Prospective Multicenter Cohort Study
Brief Title: Kasai Portoenterostomy Timing and Outcomes in Biliary Atresia
Status: Completed | Type: Observational
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Yijiang Han/Han Yijiang, Attending Physician, The Children's Hospital of Zhejiang University School of Medicine
Other Study IDs: CHZJU2025IIT013
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia | interventions — Portoenterostomy, Hepatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- ≤28 days: This observational cohort consists of infants diagnosed with type III biliary atresia who receive Kasai portoenterostomy within the first 28 days of life. Group assignment is based solely on the actual age at surgery.
  Interventions: Procedure: Kasai portoenterostomy
- 29-60 days: This observational cohort consists of infants diagnosed with type III biliary atresia who receive Kasai portoenterostomy between 29 and 60 days of life. This is a naturalistic grouping based on real-world surgical timing.
  Interventions: Procedure: Kasai portoenterostomy
- 61-90 days: This observational cohort consists of infants diagnosed with type III biliary atresia who receive Kasai portoenterostomy between 61 and 90 days of life. The cohort is defined by the exposure variable (surgical age) for comparative analysis.
  Interventions: Procedure: Kasai portoenterostomy
- 91-120 days: This observational cohort consists of infants diagnosed with type III biliary atresia who receive Kasai portoenterostomy between 91 and 120 days of life. This group represents the latest surgical timing within the study protocol.
  Interventions: Procedure: Kasai portoenterostomy

INTERVENTIONS:
Procedure: Kasai portoenterostomy — All participants in this observational study receive the standard-of-care surgical procedure, Kasai portoenterostomy (KPE). There is no study-specific intervention. The sole factor that distinguishes the four study cohorts is the natural timing of this standard surgery in the clinical course, which serves as the exposure variable for comparison. The cohorts are defined as follows:
  Cohort 1: KPE performed at or before 28 days of age.
  Cohort 2: KPE performed between 29 and 60 days of age.
  Cohort 3: KPE performed between 61 and 90 days of age.
  Cohort 4: KPE performed between 91 and 120 days of age. Participants are grouped based on their actual age at surgery in real-world practice. The study aims to compare long-term outcomes across these pre-defined surgical timing strata.

SUMMARY:
What is this study about? This study aims to find out the best timing for a major surgery called Kasai portoenterostomy (Kasai surgery) in infants with a liver disease called biliary atresia. The investigators want to see if having the surgery earlier leads to better long-term health for the baby's own liver.

Why is this important? Doctors know that early surgery is important, but it's unclear exactly how early is best. Some babies have surgery within the first month, others within 2-3 months. The investigators want to carefully compare different time windows to see which one gives the child the best chance to keep their own liver healthy and avoid a liver transplant.

How will the study work?

This is an observational study. The investigators will not change the treatment any child receives. The investigators will enroll about 200 infants from 4-5 children's hospitals in China. The investigators will simply group the infants based on their actual age at surgery:

Group 1: Surgery at 28 days old or younger.

Group 2: Surgery between 29 and 60 days old.

Group 3: Surgery between 61 and 90 days old.

Group 4: Surgery between 91 and 120 days old.

The investigators will then follow all children for 2 years after their surgery.

What will the investigators measure? The main thing the investigators want to see is how many children in each group are alive with their own liver working well 2 years after surgery (without needing a transplant). The investigators will also check many other health factors, like liver function tests, nutrition, growth, complications (like infections), and the costs of care.

What is the goal? The results of this study will help doctors and families make better, evidence-based decisions about the best time to perform this critical surgery for babies with biliary atresia.

ELIGIBILITY:
Inclusion Criteria:

* Infant age ≤ 120 days at the time of planned surgery.
* Diagnosis of type III biliary atresia confirmed by clinical presentation, laboratory tests (e.g., conjugated hyperbilirubinemia), and imaging studies (e.g., ultrasonography showing absent or abnormal gallbladder, triangular cord sign).
* Scheduled to undergo primary (first-time) Kasai portoenterostomy.
* Legal guardian(s) able to understand and provide written informed consent.

Exclusion Criteria:

* Presence of other severe congenital malformations that significantly impact prognosis or surgical risk (e.g., complex congenital heart disease requiring intervention, syndromic biliary atresia as part of a polymalformation complex).
* Pre-existing evidence of decompensated cirrhosis (e.g., refractory ascites, hepatopulmonary syndrome, or hepatic encephalopathy) prior to surgery.
* Previous history of any liver surgery (including prior Kasai portoenterostomy attempt or liver biopsy via laparotomy).
* Any condition that, in the opinion of the investigator, would make the infant unsuitable for participation or could interfere with the completion of follow-up (e.g., severe concurrent infection, life-limiting non-hepatic disease).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This prospective observational cohort study will enroll approximately 200 infants (age ≤120 days) diagnosed with type III biliary atresia (BA) who are scheduled to undergo their first (primary) Kasai portoenterostomy (KPE). Participants will be recruited from 4-5 pediatric tertiary care centers in China. Enrollment is based on real-world clinical presentation and surgical planning; no study-specific intervention is administered. Infants will be grouped into four natural cohorts according to their actual age at surgery: ≤28 days, 29-60 days, 61-90 days, and 91-120 days. The population will be followed prospectively for 24 months postoperatively to compare long-term outcomes across these surgical timing strata.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2025-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Native Liver Survival Rate | 24 months after Kasai surgery
  Percentage of participants alive without liver transplantation at 24 months post-operation.

SECONDARY OUTCOMES:
Clearance of Jaundice | At 3 months and 6 months after surgery
  Proportion of participants achieving serum total bilirubin <20 μmol/L.
Incidence of Postoperative Cholangitis | Within 24 months after surgery
  Proportion of participants experiencing ≥1 episode of cholangitis.
Incidence of Portal Hypertension | Within 24 months after surgery
  Proportion diagnosed with portal hypertension.
Longitudinal Change in Liver Enzymes | Preop, 2 weeks, 1, 3, 6, 12, 18, 24 months postop
  Trajectory of liver enzyme levels.
Change in Weight-for-Age Z-score (WAZ) | Preop, 6, 12, 24 months postop
  Change in weight-for-age Z-score.
Perioperative Complication Rate | Within 30 days after surgery
  Proportion with any complication.

OTHER OUTCOMES:
Direct Medical Costs of BA Management | From surgery hospitalization until 24 months postop
  Total direct medical costs.
Longitudinal Change in Serum 25-Hydroxyvitamin D Level | Preop, 6, 12, 24 months postop
  Change in 25(OH)D concentration.
BA-Related Re-hospitalization Rate | Within 24 months after surgery
  Proportion re-hospitalized.
Postoperative Hospital Length of Stay | From surgery to first discharge, assessed up to 60 days
  Postoperative Hospital Length of Stay
Duration of Kasai Portoenterostomy | On the day of surgery
  Total operative time.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, China